CLINICAL TRIAL: NCT05019469
Title: Investigating Responsive Vibration Cueing Modalities From a Wearable Device to Overcome Gait Freezing in Parkinson's Disease
Brief Title: Overcoming Gait Freeze in Parkinson's Disease Using Responsive Cueing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS_216723; 18/SW/0235 (Other: NHS Health Research Authority REC)
Record Dates: First submitted 2021-08-04; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Gait freezing; Cueing; Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm of study (Experimental): Single Arm. During each study session the participant undertakes 4 walking/activity circuits. During each circuit the participant receives either continuous cueing, responsive cueing (delivered in response to gait freezing), no cueing and no device. The ordering of the interventions/circuits are systematically alternated for each participant.
  Interventions: Device: Rhythmic vibration cueing (lower leg)

INTERVENTIONS:
Device: Rhythmic vibration cueing (lower leg) — A non-invasive wearable device worn against both gastrocnemius muscles provides rhythmic vibrations when triggered.

SUMMARY:
The aim of this pilot/feasibility study is to test if delivering rhythmic vibration cues to the lower legs, specifically in response to gait defects (rather than continuously), can improve walking quality and overcome gait freezing in Parkinson's disease.

During the study, people with Parkinson's disease that suffer from regular (daily) gait freezing will undertake a series of walking/activity circuits, receiving continuous cueing, responsive cueing (delivered in response to gait freezing), no cueing and no device. Vibration cueing is provided by a non-invasive wearable device prototyped at the University of Oxford, worn on the lower legs during 3 circuits. A series of walking metrics will be analysed.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive, neurodegenerative disorder that impairs the ability to control movement. Gait freezing is an inability to walk spontaneously and continuously, and affects nearly half of PD patients, reducing quality of life and contributing to increased fall risk. Cueing (with visual, auditory or somatosensory stimuli) is an effective way to improve walking quality in people with PD. In this pilot study we aim to test if delivering rhythmic vibration cues acutely, specifically in response to gait defects, can improve walking quality and overcome gait freezing in PD.

During the study, people with PD that suffer from regular (daily) gait freezing, but who are able to stand and walk with minimal assistance, undertake 4 walking/activity circuits. During each of the circuits participants receive either continuous cueing, responsive cueing (delivered in response to gait freezing), no cueing and no device. Cueing is provided by a non-invasive wearable movement-tracking cueing device prototyped at the University of Oxford (approximately the size of a smart phone), worn on the lower legs during 3 circuits. The ordering of the interventions/circuits are systematically alternated for each participant. The impact of responsive cueing on walking ability can be determined by analysis of walking metrics across the circuits.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participant is fluent in English.
* Participant is aged 18-90 years inclusive
* Patients in whom the clinical diagnosis is stated as idiopathic Parkinson's disease or Parkinson's disease (PD).
* Participant self-reports a history of daily gait freezing (several times a day), but should be able to stand and walk freely for short periods with minimal assistance.
* Participant has no evidence for significant cognitive impairment.
* In the investigator's opinion, is willing and able to comply with all trial requirements.

Exclusion Criteria:

* Participant has a medical or psychiatric illness that would interfere with completing initial and follow up assessments.
* Participant has severe mental impairment, dementia or psychosis determined either by a prior diagnosis by a medical professional with relevant expertise, or by subjective assessment by the research team during the pre-study questionnaire (e.g. an inability to comprehend questions).
* Active participation in a clinical drug trial.
* Female who is pregnant, lactating or planning pregnancy during the course of the investigation. This information will be provided to us by the patient during recruitment screening.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Patients with frequent (daily) falls at home or out of home, or who demonstrate a high fall risk during the study.
* Patients with atypical parkinsonism (eg MSA, PSP, CBD).
* Patients who have had Deep Brain Stimulation for their PD.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Step frequency | Data collected during 1 hour sessions up to study completion.
  The primary objective is to test if gait-freeze initiated vibration cues, provided at the lower-leg, can improve gait/walking quality in PD patients. The primary outcome measure will be cadence (step frequency) with other gait measurements including frequency and duration of gait freeze events, continuous walking time, left/right rhythm and stride length. Measurements extracted from video data collected during 1 hour study sessions. Change in these measurements assessed between cued (intervention) and no-cue (no intervention) walking circuits for each participant.

SECONDARY OUTCOMES:
Automated gait freeze detection | Movement data collected during 1 hour sessions up to study completion.
  Generation of algorithms capable of recognising gait freeze events from device movement data with >80% accuracy. Algorithm development to identify changes in accelerometer (g) and gyroscope (rsp) data from leg-worn devices indicative of gait freeze events. Algorithm accuracy expressed as % sensitivity and % specificity for identifying gait freeze events from movement data relative to observer time stamps.

CONTACTS AND LOCATIONS:
Overall Officials: James Cantley, PhD, Principal Investigator — University of Oxford
Locations (1):
- The Bosworth Clinic, Cassington, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data points will be shown in the manuscript/publication reporting the study outcomes.